CLINICAL TRIAL: NCT06829953
Title: Geospatial and Ecological Momentary Assessment Technology and Activity Engagement for At-risk Youth (Get ActivE)
Brief Title: Get ActivE Study for At-risk Youth
Acronym: GetActivE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Children's Hospital of Philadelphia (Other); University of Oregon (Other); National Institute of Mental Health (NIMH) (NIH); Columbia University (Other)
Responsible Party: Principal Investigator, Jamie Zelazny, Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY22040034; P50MH115838 (NIH)
Record Dates: First submitted 2025-02-11; First posted 2025-02-17 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Anhedonia; Depression and Suicide Ideation
Keywords: Behavioral Activation; Health Coach; Anhedonia; Minority Youth; Suicide
MeSH Terms: conditions — Anhedonia; Depression; Suicide | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Examination of implementation outcomes, target engagement, and preliminary effectiveness of GET ActivE via a randomized trial with 75 adolescents (age 12-18, 35% Black, 10% Hispanic) at risk for suicide (moderate-severe depression) and with difficulties with anhedonic symptoms identified in primary care.
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor will be blinded to the randomized treatment arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Activity Monitoring Alone (Active Comparator): Participants who are eligible for the GET Active Study and are randomly assigned to Treatment As Usual will be asked to download a mobile sensing activity monitoring app called the Effortless Assessment of Risk States (EARS) app which will derive activity data. The activity data will be collated to yield weekly summary measures that will be sent via short messaging services (SMS) text messaging to participants randomized to the control condition for viewing.
  Interventions: Behavioral: Treatment As Usual
- GET ActivE (Experimental): GET ActivE intervention uses the Vira mobile application and a health coach, integrating mobile sensing, self-report assessment, and just-in-time nudges and notifications from a health coach to increase patient activity and promote positive mood cycles. A health coach reinforces Behavioral Activation (BA) principles and encourages engagement with activities by composing and triggering appropriate intervention nudges and messages (by text, phone call, video call, chat, email, etc.) specific to activity patterns and mood ratings highlighted on the Vira app. The health coach reviews the patient's data from the Vira practitioner dashboard and will follow up with patients at least weekly (and caregivers periodically) to reinforce behaviors that are consistent with BA and personally relevant based on the participant's own mobile sensing data and mood ratings.
  Interventions: Behavioral: GET ActivE

INTERVENTIONS:
Behavioral: GET ActivE — The GET ActivE health coach will review data from the Vira app and send nudges to the participant with insights encouraging them to engage in activities that bring enjoyment or pleasure.
  Arms: GET ActivE
Behavioral: Treatment As Usual — Participants randomized to Treatment As Usual may have access to activity data from an app and receive summary information about activity patterns at the end of their participation.
  Arms: Activity Monitoring Alone

SUMMARY:
The study will adapt and deploy a digital Behavioral Activation app with mobile sensing, supported by health coaches, that encourages youth to engage in positive activities. The study has the potential to offer a low-cost and scalable behavioral intervention that may decrease risk of suicide among at-risk youth. This research will examine specifically whether an intervention involving an app called Vira, combined with health coaching (GET ActivE) can improve enjoyment for teens coping with depression. Research participants will be randomly assigned to one of two study intervention. One study intervention involves a) downloading an app called Vira and engaging by responding to a daily question, and b) participating in a conversation via text, phone, or messages through an appt with a health coach. The health coach will use the Vira app and principles from evidence-based therapy and behavior change to provide users with insights to sustain well-being and better manage risk factors for suicidal thoughts and behaviors such as depressed mood and behavioral withdrawal. The second study intervention involves downloading an app called EARS and responding to a daily question.

DETAILED DESCRIPTION:
Aim 3 (Randomized Pilot): To examine implementation outcomes, initial effectiveness, and equity across outcomes in a pilot randomized trial (n=75, 2:1 randomization, 35% Black, 10% Hispanic) of GET ActivE vs. Activity Monitoring Alone. H3a. The study will observe high GET ActivE feasibility (50% of eligible youth approached will enroll; completion >50%; attrition <20%; response to health coach contacts >80%); acceptability (>80%); and appropriateness (>80%). H3b. Youth who receive GET ActivE will show greater improvement in anhedonia (primary outcome) and H3c. depression severity and suicidal risk (secondary outcomes). H3d. Outcomes will be equitable by race. H3e. Exploratory (mechanistic): GET ActivE will lead to decreased depression and suicidal risk through increased activity and reward responsiveness.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents age 12-18
* Current moderate to severe depression (PHQ-9-M > 11)
* Current clinically significant anhedonia, operationalized as PHQ-9-M anhedonia item score > 1
* English language fluency and literacy level sufficient to engage in study protocol
* Willing to download the app on their smart phones

Exclusion Criteria:

* Evidence of mania, psychosis, or developmental disability precluding comprehension of study procedures per electronic health record review and phone screen.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-03-27 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
GET ActivE Feasibility | 3 months
  The study will observe high GET ActivE intervention feasibility (50% of eligible youth approached will enroll; completion >50%; attrition <20%)
Response to Health coach contacts | 3 months
  Participants will respond to health coach contacts >80%
GET ActivE Acceptability | Post intervention follow up; up to 3 months
  Acceptability of the GET ActivE intervention will be assessed through the 4 item Acceptability of Intervention Measure (AIM). Individual item scores are summed. Scale values range from 1 to 5. No items are reverse scored. Higher scores indicate greater acceptability. The items include questions to determine if intervention is appealing to, liked by, welcomed by, and approved by study population.
GET ActivE Appropriateness | Post intervention follow up; up to 3 months
  Intervention appropriateness of the GET ActivE intervention will be assessed through 4 item Intervention Appropriateness Measure (IAM). Individual item scores are summed. Scale values range from 1 to 5. No items are reverse scored. Higher scores indicate greater appropriateness. The items include questions to determine if intervention is a good match, fitting, suitable, or seems applicable to the study population.

SECONDARY OUTCOMES:
Anhedonia | baseline and follow up timepoints 1 month, 3 months, 6 months, 12 months
  Anhedonia will be assessed using the self-reported Behavioral Avoidance/Inhibition (BIS/BAS), 24 item scale. The scoring ranges from 1-4 and response options include: Very true for me (1); somewhat true for me (2); somewhat false for me (3); very false for me (4). Total range of scores possible is 24-96. The lower the score reported on BIS/BAS, the less pleasure or enjoyment a responder feels and more anhedonic symptoms are expressed.

OTHER OUTCOMES:
Suicidal thoughts and behaviors | baseline and follow up timepoints 1 month, 3 months, 6 months, 12 months
  Suicidal attempt & ideation will be measured through the Columbia Suicide Severity Rating Scale (C-SSRS). Assign score of 0 if no ideation/behavior present and assign a score of 1 if ideation/behavior present. A "yes" answer any time during treatment to any 1 of the 5 suicidal behavior questions (Categories 7-10) on the C-SSRS. C-SSRS Categories 7-10 are as follows: 7-Aborted Attempt 8-Interrupted Attempt 9-Actual Attempt (non-fatal) 10-Completed Suicide. Any score greater than 0 is important/may indicate need for intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Zelazny, PhD, MPH, RN, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Consistent with the NIMH's data sharing and data use policies this research study and clinical trial will be compliant with requirements for depositing data with the NIMH Data Archive (NDA) in the National Database for Clinical Trials Related to Mental Illness (NDCT). Specific statements will be added to the consent forms to allow for data sharing. The final completely de-identified dataset(s) will include demographic and clinical data at baseline, and primary and secondary outcomes for all studies.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Individual participant data will be available in a deidentified manner through the NIMH Data Archive indefinitely.
Access Criteria: Verified researchers may request the data through the NIMH Data Archive.